CLINICAL TRIAL: NCT04334109
Title: Comparative Effectiveness of Family DSMES and Standard DSMES Among Diverse Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 260059
Record Dates: First submitted 2020-03-26; First posted 2020-04-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-DSME (Experimental): Approach
  * Family motivational interviewing techniques
  * Family goal setting
  * Understanding supportive and nonsupportive family behaviors
  * Family behavioral changes Mode of Delivery
  * Group sessions delivered by a certified diabetes educator (CDE) to patients and their family members Dosage
  * 10 hours delivered in one-hour sessions over 10 weeks Participants
  * 300 patients with T2D and 300 family members (family members will take part in educational sessions and data collection)
  Interventions: Behavioral: Family Diabetes Self-Management Education and Support
- Standard-DSME (Active Comparator): Approach
  * Individual motivational interviewing techniques
  * Individual goal setting
  * Individual behavioral changes Mode of Delivery
  * Group sessions delivered by a CDE to patients Dosage
  * 10 hours delivered in one-hour sessions over 10 weeks Participants
  * 300 patients with T2D (family members will take part in data collection but not educational sessions)
  Interventions: Behavioral: Standard Diabetes Self-Management Education and Support

INTERVENTIONS:
Behavioral: Family Diabetes Self-Management Education and Support — Family Diabetes Self-Management Education and Support demonstrates the effectiveness of family-centered models of DSME that explicitly address diabetes self-management within a family context by educating both patients and family members and focusing on family motivational interviewing, family goal setting, understanding supportive and nonsupportive behaviors, and family behavioral changes.
  Arms: Family-DSME
Behavioral: Standard Diabetes Self-Management Education and Support — Diabetes Self-Management Education and Support demonstrates the effectiveness of individual model DSMES that explicitly address diabetes self-management within an individual context by educating individual patients on individual motivational interviewing, individual goal setting, and individual behavioral changes.
  Arms: Standard-DSME

SUMMARY:
The investigators will conduct a fully-powered, comparative effectiveness randomized controlled trial that includes up to 600 patients with type 2 diabetes (T2D) and 600 of their family members. Patients with T2D will be randomly assigned to either the Family-DSMES arm or the Standard-DSMES arm, with 300 patients in each arm. In the Family-DSMES arm, one of each patient's family members will take part in the educational sessions (family members defined below). Baseline and follow-up data (immediate post-intervention, 6 months post-intervention, and 12 months post-intervention) will be collected from patients and family members in both study arms. In the Standard-DSMES arm, data will be collected from family members, but they will not participate in educational sessions. In both arms, the investigators will obtain a medical records release to abstract outcomes at 18 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years of age
* have T2D (HbA1c ≥ 7.0)
* speak English
* a family member willing to take part in the study

Exclusion Criteria:

* have received formal DSME in the past three years
* have a condition that makes it unlikely for them to be able to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Change in mean HbA1c (NGSP%) from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  A Siemens analyzer will be utilized to calculate HbA1c (%) for each participant at every time point (except for 18 months post-intervention, which will be collected through medical record abstractions). Changes in the primary outcome measure will be assessed from baseline to each follow-up time point. The primary analytic approach will use general linear models, including mixed effects linear regression models for continuous repeated measures, to model the mean outcome difference and covariance structures between the treatment arms. Analyses will be adjusted for baseline differences in demographic, socioeconomic, and clinical variables, all within repeated mixed linear regression models. Clustering effects within the intervention delivery groups (i.e., within the DSMES classes) will be accounted for in the model as a random effect. We will adjust for potential clinic variations as a dummy coded variable in our model.

SECONDARY OUTCOMES:
Change in mean BMI from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  BMI will be collected by measuring participant height (without shoes) using a stadiometer, and measuring participant weight (without shoes) using a calibrated digital scale. Weight and height will be used to compute a continuous measure of BMI. BMI at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean waist circumference from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention medical record abstraction | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Waist circumference will be collected by measuring participant's waist using a flexible tape measure. Waist circumference at 18 months post-intervention will be abstracted from participant medical records.The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean blood pressure (systolic & diastolic, mmHg) from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Blood pressure will be measured with a sphygmomanometer and stethoscope or digital blood pressure device with the participant seated and arm elevated. Blood pressure at 18 months post-intervention will be abstracted from participant medical records.The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean total cholesterol (mg/dL) from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention medical records abstraction
  Through finger prick blood collection, point of care tests will be used used to test lipids using a commercial lipid panel kit and Cholestech LDX analyzer. Total cholesterol at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean high-density lipoproteins (HDL) from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Through finger prick blood collection, point of care tests will be used used to test HDL using a commercial lipid panel kit and Cholestech LDX analyzer. HDL at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean low-density lipoproteins (LDL) from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Through finger prick blood collection, point of care tests will be used used to test HDL using a commercial lipid panel kit and Cholestech LDX analyzer. LDL Blood pressure at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean triglycerides from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Through finger prick blood collection, point of care tests will be used used to test triglycerides using a commercial lipid panel kit and Cholestech LDX analyzer. Triglycerides at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in mean blood glucose from baseline to immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Through finger prick blood collection, point of care tests will be used used to test random blood glucose (not fasting). Blood glucose at 18 months post-intervention will be abstracted from participant medical records. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in diabetes self-management behaviors from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention
  The Summary of Diabetes Self-Care Activities (SDSCA) will be used to measure engagement in self-management activities. The SDSCA consists of 12 items to assess the self-reported frequency of performing diabetes self-care tasks, including testing blood sugar, following healthful eating plans, and exercising regularly. The SDSCA will be administered to participants at baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in diabetes self-efficacy from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention
  The Diabetes Management Self-Efficacy Scale (DMSES) will be used to measure patient's confidence in managing their diabetes. The DMSES consists of 20 items to assess self-reported confidence in managing aspects of their diabetes. The DMSES will be administered to participants at baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in medication adherence from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention
  The Adherence to Refills and Medications Scale for Diabetes Medicines (ARMS-D) will be used to measure patient's adherence to their medications (if prescribed). The ARMS-D consists of 11 items to assess self-reported adherence to diabetes medications. The ARMS-D will be administered to participants at baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in diabetes-related distress from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention
  The Problem Areas in Diabetes Scale (PAID)-5 will be used to measure diabetes distress. The PAID-5 consists of 5 items to assess self-reported diabetes-related emotional distress, including feeling scared or depressed. The PAID-5 will be administered to participants at baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.
Change in diabetes-related quality of life from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention | Baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention
  The DAWN2 Impact of Diabetes Profile (DIDP) will be used to measure the perceived impact of diabetes on patients' quality of life. The DIDP consists of 6 items to assess self-reported impacts on quality of life, including physical health, financial situation, and relationships with others. The DIDP will be administered to participants at baseline, immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. The analytic approach for secondary outcomes will be similar to those used for the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayberry LS, Felix HC, Hudson J, Curran GM, Long CR, Selig JP, Carleton A, Baig A, Warshaw H, Peyrot M, McElfish PA. Effectiveness-implementation trial comparing a family model of diabetes self-management education and support with a standard model. Contemp Clin Trials. 2022 Oct;121:106921. doi: 10.1016/j.cct.2022.106921. Epub 2022 Sep 9. PMID 36096282